CLINICAL TRIAL: NCT01294930
Title: Indicators of Operative and Postoperative Complications in Patients Operated for Hip Fracture
Acronym: IOPC
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Vrinnevi Hospital (Other)
Responsible Party: Principal Investigator, Joachim Zdolsek, MD, PhD, University Hospital, Linkoeping
Other Study IDs: IOPC
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Hip Fracture
Keywords: hip fracture; mortality; complications
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hip fracture: Patients operated for hip fracture, giving informed consent
  Interventions: Other: Urine density

INTERVENTIONS:
Other: Urine density — measurement of urine color, density and plethysmographic variability index before and during surgery.
  Other Names: - Urine color; - Urine density; - Plethysmographic variabilty

SUMMARY:
Patients operated for hip fractures are older and have several conditions that have negative influences on the perioperative and postoperative prognosis.

Hip fractures can also be painful, which is stressful for the physiology of the patient. Many old patients have received to little fluid intake. They often have diuretic therapy, which even worsens dehydration/hypovolemia.

Some patients have to wait several days for surgery. Several studies have shown a high degree of complications and an increased mortality in this patient group.

Early preoperative optimization can improve the outcome. The available methods for optimization of the patient are complicated and time consuming.

The investigators wish with this study to try new approaches to find which patients still are dehydrated when they come to the operation ward.

The aim is to measure the color and density of the urine as well as to register the the variability in the plethysmographic curve before spinal anaesthesia.

These results will be compared to circulatory instability during and after surgery as well as to postoperative complications.

DETAILED DESCRIPTION:
All patients with hip fractures planed fore surgery at the Hospital in Norrkoping will come into consideration to participate in study.

Many will however not be able to give consent. These will not be included in the study.

Directly preoperatively urine will be collected. Color and density will be measured/registered.

The pulseoximeter reading will be registered (Saturation, pulse, PI and PVI) before spinal anaesthesia and after spinal anaesthesia as well as during the surgery.

Two to three days postoperatively a follow up will be performed, to register complications (Circulatory instability, confusion, infection, affected kidney function/creatinine rise).

30 day postoperative mortality will also be controlled.

These results will be compared, to see if pulse oximeter readings or urine concentration can predict complications.

ELIGIBILITY:
Inclusion Criteria:

* patients with hip fracture
* operation for the hip fracture
* informed consent

Exclusion Criteria:

* patients not giving consent
* patients not being able to understand information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hip fracture operated at the hospital in Norrkoeping
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
mortality | 30 days
  30-day mortality related to indices of dehydration (urine and pulse oximetry)

SECONDARY OUTCOMES:
operative and postoperative complications | 3 days
  Number of complications according to a prospective list

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hahn, MD PhD Prof, Study Director — University Hospital, Linkoeping
Locations (1):
- Anaesthesia dept, Vrinnevisjukhuset, Norrköping, Norrkoeping, Sweden

REFERENCES:
- [Derived] Ylinenvaara SI, Elisson O, Berg K, Zdolsek JH, Krook H, Hahn RG. Preoperative urine-specific gravity and the incidence of complications after hip fracture surgery: A prospective, observational study. Eur J Anaesthesiol. 2014 Feb;31(2):85-90. doi: 10.1097/01.EJA.0000435057.72303.0e. PMID 24145802